CLINICAL TRIAL: NCT00867815
Title: Prospective Case Crossover Study to Assess Whether PDE5 Inhibitor Exposure in Men Increases the Risk for the Development of Non-arteritic Anterior Ischemic Optic Neuropathy (NAION)
Brief Title: PDE5 Inhibitor Use and Non-arteritic Anterior Ischemic Optic Neuropathy (NAION)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 12912; 2010-023586-22 (EudraCT Number)
Record Dates: First submitted 2009-03-23; First posted 2009-03-24 (Estimated); Results first posted 2019-01-23 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Anterior Ischemic Optic Neuropathy
Keywords: Non-arteritic Anterior Ischemic Optic Neuropathy; NAION; PDE5 inhibitors; vardenafil; Levitra; sildenafil; Viagra; Tadalafil; Cialis; acute vision loss; vision loss; blurred vision; optic neuropathy; erectile dysfunction.
MeSH Terms: conditions — Optic Neuropathy, Ischemic; Blindness; Vision Disorders; Optic Nerve Diseases; Erectile Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Drug: Diagnostic procedures

INTERVENTIONS:
Drug: Diagnostic procedures — The patients will not receive any study drug in this study. The patients will have ophthalmological (eye) examinations, blood work and will complete an interview

SUMMARY:
The primary objective of this study is to determine whether the use of PDE5 inhibitors (vardenafil, sildenafil, or tadalafil) increases the risk for the development of NAION.

DETAILED DESCRIPTION:
Collected data will be compared to historic data of the same participant in case-crossover design.

ELIGIBILITY:
Inclusion Criteria:

* NAION onset within 45 days before entry to the study
* NAION onset definable by the subject within a 2 calendar day window
* Men who have taken at least 1 dose of PDE5 inhibitor(s) at any time in the 1 year prior to enrollment in the study
* Age 40 years or older

Exclusion Criteria:

* History of multiple sclerosis or optic neuritis
* Evidence of temporal arteritis
* History of vasculitis or collagen vascular disease
* Previous history of NAION

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-07-13 (Actual); Primary Completion 2017-12-29 (Actual); Study Completion 2018-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (13):
- United States (11):
  - Greider Eye Associates, Vista, California
  - Palm Beach Eye Center, Atlantis, Florida
  - West Coast Eye Care, Fort Myers, Florida
  - National Ophthalmic Research Institute, Fort Myers, Florida
  - Sarasota Retina Institute, Sarasota, Florida
  - Midwest Eye Institute, Indianapolis, Indiana
  - Spoor and Associates, Warren, Michigan
  - Asheville Eye Associates, Asheville, North Carolina
  - Office of Dr. Avrom Epstein, MD, Columbus, Ohio
  - Tulsa Clinical Research, LLC, Tulsa, Oklahoma
  - Retinal and Ophthalmic Consultants, Houston, Texas
- Save Sight Institute, Sydney, New South Wales, Australia
- Midwest Eye Institute, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started on 13 JUL 2009 (FPFV) and the date of last visit was 29 DEC 2017 (LPLV).
Pre-assignment Details: There were 10 screening failures. The primary reasons for screen failure are protocol violation (8 participants) and consent withdrawn (2 participants)
Groups:
- PDE5 Inhibitor Use & Risk of NAION: Participants were assessed at 2 visits. Visit 1 (Day 1) included screening, confirmation of the diagnosis of NAION, enrollment, and collection of data on PDE5 inhibitor and other concomitant medication use. Visit 2 (Day 90+/-30) was a follow-up visit to document the persistence of vision loss and confirm the diagnosis of NAION. No interventional treatment was administered in the context of this study.
Period: Overall Study
Arm/Group | PDE5 Inhibitor Use & Risk of NAION
Started (Safety Analysis Set) | 10
Completed | 9
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | PDE5 Inhibitor Use & Risk of NAION
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Confirmed Diagnosis of Non-arteritic Anterior Ischemic Optic Neuropathy (NAION)
Description: The study population consisted of adult men, first diagnosed with NAION which started within 45 days before study start and took PDE5 inhibitors (vardenafil, sildenafil, tadalafil or avanafil) in the 1 year prior to enrollment.
Time Frame: Up to 45 days prior to study enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | PDE5 Inhibitor Use & Risk of NAION
Number analyzed (Participants) | 10
Participants | 10

2. Secondary Outcome: Number of Participants With Most Frequent Medical History Findings by Primary System Organ Class at Visit 1
Description: The safety population includes participants who signed informed consent and who had any of the following collected at Visit 1 for safety: laboratory values, physical exam, any eye exams, or adverse events.
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | PDE5 Inhibitor Use & Risk of NAION
Number analyzed (Participants) | 10
Participants
  Metabolism and nutrition disorders | 7
  Eye disorders | 6

3. Secondary Outcome: Number of Participants With Any Adverse Events Reported at Visit 2
Description: An adverse event is any untoward medical occurrence in a subject or clinical investigation subject and can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally occurring during the trial.
Time Frame: From informed consent signed up to Visit 2 (Day 90+/-30)
Measure: Count of Participants; unit: Participants
Arm/Group | PDE5 Inhibitor Use & Risk of NAION
Number analyzed (Participants) | 10
Participants | 3

ADVERSE EVENTS:
Time Frame: From inform consent signed up to approximately 3 months after first diagnosis of NAION
Arm/Group | PDE5 Inhibitor Use & Risk of NAION
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 2/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PDE5 Inhibitor Use & Risk of NAION (N=10)
Optic ischaemic neuropathy (Eye disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PDE5 Inhibitor Use & Risk of NAION (N=10)
Eye irritation (Eye disorders) | 1 (1)
Ocular discomfort (Eye disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Study was prematurely terminated, hence no statistical analysis was performed due to small sample of population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The agreed point of publication is 12-18 months after database lock at the earliest.

* Bayer will have up to 30/45 days to review publications, and may request an additional publication delay of up to 60 days to allow for filing a Patent Application (if applicable).
* No publication of single center data should be done prior of publication if multi -center data)。

DOCUMENTS (2):
  • Study Protocol (2016-03-02): https://cdn.clinicaltrials.gov/large-docs/15/NCT00867815/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-20): https://cdn.clinicaltrials.gov/large-docs/15/NCT00867815/SAP_001.pdf